CLINICAL TRIAL: NCT01431365
Title: Does an Acute Bout of Exercise Affect Smoking Topography?
Brief Title: Effect of an Acute Bout of Exercise on Smoking Topography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Harry Prapavessis, Dr., University of Western Ontario, Canada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SmokingTopography210
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Cancer
Keywords: exercise; topography; cravings; smoking behaviour
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate Exercise Group (Experimental): The moderate exercise condition will involve participants walking briskly (equivalent to moderate intensity) on a treadmill for 10 minutes. Moderate intensity exercise will be defined as 40-68% of the resting heart rate reserve. Heart rate (HR) will be monitored in participants using a Polar RS100 Heart Rate monitor to serve as a guide for participants to attain the appropriate intensity.
  Interventions: Behavioral: Moderate Exercise Group
- Passive Sitting Group (Active Comparator): The passive sitting condition will involve participants sitting passively for 10 minutes on a chair. Heart rate (HR) will be monitored in participants of the passive sitting group to help maintain group equivalency (with the moderate exercise condition) in regards to distraction effects and researcher contact.
  Interventions: Behavioral: Passive Sitting Group

INTERVENTIONS:
Behavioral: Moderate Exercise Group — Participants will be required to walk briskly (equivalent to moderate intensity) on a treadmill for 10 minutes.
  Other Names: Physical activity
  Arms: Moderate Exercise Group
Behavioral: Passive Sitting Group — Participants will be required to sit passively for 10 minutes on a chair.
  Other Names: Sedentary
  Arms: Passive Sitting Group

SUMMARY:
Smokers will complete questionnaires and smoking behaviour will be examined. After abstaining from smoking for approximately 18 hours, they will be randomized to a moderate intensity exercise group or passive sitting group. Smoking behaviour (time to first puff) will be assessed following treatment.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death in Canadians (Canadian Cancer Society, in which cigarette smoking is responsible for 85% of these cases. Smoking topography, a key facet of smoking behaviour, can be subjectively or objectively measured by quantifying puff volume, maximum puff velocity, interpuff interval, puff duration, number of puffs per cigarette, and the time to smoke a single cigarette. Smoking topography can estimate exposure to carcinogenic toxins present in cigarette smoking (Djordjevic, Hoffman, & Hoffman, 1997). Evidence exists to support that exercise modifies smoking topography (Katomeri & Taylor 2006; Mikhail, 1983; Reeser, 1983; Zacny & Stitzer, 1985).

Recently, Faulkner and colleagues (2011; N = 18) were the first to implement a handheld smoking topography device (CReSS Pocket) to measure smoking behaviour in the context of an acute bout of exercise after a temporary period of abstinence. They found that brisk walking influences an individual's smoking topography. In specific, participants assigned to the exercise condition smoked less per puff and took shorter puff durations, compared to the passive sitting condition. Overall, smoking topographical studies require further investigation due to methodological flaws in order to allow for the objective collection of smoking behaviour data and improved external validity in a sufficiently powered study. Furthermore, the role of cravings, withdrawal and affect as potential mediators of topographical changes due to exercise is a novel area of research.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 64 years of age
* Smoke 10 cigarettes or more per day
* Not have any medical condition that is contraindicative for exercise
* Not be pregnant or intending on being pregnant over the course of the study
* Be able to read and write in English
* Have a telephone or an email account so that they can be contacted
* Completed the Physical Activity Readiness Questionnaire (PAR-Q)
* Have Medical Doctor's clearance if they answer "YES" to one or more questions on the Physical Activity Readiness Questionnaire (PAR-Q)
* Have not been engaged in a serious quit attempt in the last six months
* Have been smoking for more than 2 years
* Must not be suffering from an illness (e.g. cold) that would affect their typical smoking behaviour

Exclusion Criteria:

* Contraindication to exercise (e.g., disability, unstable angina)
* On medication for physical and/or mental health reasons that would make compliance with the study protocol difficult or dangerous
* Have substance dependency problems (e.g., alcohol)
* Are pregnant
* Be younger than 18 years of age
* Be 64 years or older prior to completion of the study
* Have been engaged in a serious quit attempt in the last six months
* Have been smoking for less than 2 years
* Suffering from an illness (e.g. cold) that would affect their typical smoking behaviour

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Smoking topography | One week
  Smoking topography will be assessed using the Clinical Research Support System (CReSS) Pocket, a computer-based, battery-powered, hand-held unit by Plowshare Technologies®. The CReSS Pocket has an orifice flow meter mouthpiece, and a pressure drop related to the flow rate that is produced when a puff is taken. From the flow rate, the CReSS derives puff count (number of puffs per cigarette), puff volume (the volume of carbon monoxide take in during each puff), puff duration (length of time for each puff), inter-puff interval (amount of time between puffs), and time to first puff.

SECONDARY OUTCOMES:
Withdrawal symptoms | One week
  Changes in cravings, positive and negative affect, and mood and physical symptoms will be assessed using three questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Prapavessis, Ph.D., Principal Investigator — Western University, Canada
Locations (1):
- Exercise and Health Psychology Laboratory- University of Western Ontario, London, Ontario, Canada

REFERENCES:
- [Background] Aveyard P, West R. Managing smoking cessation. BMJ. 2007 Jul 7;335(7609):37-41. doi: 10.1136/bmj.39252.591806.47. No abstract available. PMID 17615224
- [Background] Ussher MH, Taylor A, Faulkner G. Exercise interventions for smoking cessation. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD002295. doi: 10.1002/14651858.CD002295.pub3. PMID 18843632
- [Background] Taylor AH, Ussher MH, Faulkner G. The acute effects of exercise on cigarette cravings, withdrawal symptoms, affect and smoking behaviour: a systematic review. Addiction. 2007 Apr;102(4):534-43. doi: 10.1111/j.1360-0443.2006.01739.x. PMID 17286639
- [Background] Taylor A, Katomeri M. Walking reduces cue-elicited cigarette cravings and withdrawal symptoms, and delays ad libitum smoking. Nicotine Tob Res. 2007 Nov;9(11):1183-90. doi: 10.1080/14622200701648896. PMID 17978993
- [Background] Zacny JP, Stitzer ML. Effects of smoke deprivation interval on puff topography. Clin Pharmacol Ther. 1985 Jul;38(1):109-15. doi: 10.1038/clpt.1985.143. PMID 4006371
- [Background] Faulkner GE, Arbour-Nicitopoulos KP, & Hsin A. Cutting down one puff at a time: The acute effects of exercise on smoking behavior. Journal of Smoking Cessation (5): 130-135, 2010.
- See also: Exercise and Health Psychology Laboratory — http://www.ehpl.uwo.ca